CLINICAL TRIAL: NCT01853969
Title: Typing Proficiency Following Carpal Tunnel Release
Status: Completed | Type: Observational
Sponsor: Vanderbilt University (Other)
Collaborators: Orthopedic Research and Education Foundation (Other)
Responsible Party: Principal Investigator, Donald Lee, Professor of Orthopaedic Surgery, Vanderbilt University
Other Study IDs: 101131
Record Dates: First submitted 2013-05-09; First posted 2013-05-15 (Estimated); Last update posted 2015-09-17 (Estimated); Status verified 2015-09

CONDITIONS: Carpal Tunnel Release

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients who have carpal tunnel release surgery
  Interventions: Other: Typing assessment

INTERVENTIONS:
Other: Typing assessment

SUMMARY:
This study will investigate how soon a patient's typing proficiency returns to their pre-operative levels following carpal tunnel release surgery. In order to determine this, patients will undergo typing tests at different time points that will record their typing accuracy and speed. The results will then be compared to determine on average how soon a person returns to their pre-operative baseline results.

DETAILED DESCRIPTION:
Carpal tunnel syndrome is a condition in which the median nerve is compressed at the wrist. It causes such symptoms as numbness, tingling, weakness, muscle damage, and pain. If non-operative treatments do not work generally patients go on to carpal tunnel release surgery in which the transverse carpal ligament is released. After surgery patients usually return to work with no restrictions within six weeks. Patients often ask how soon they are able to return to typing after surgery, and what their typing ability will be like after surgery. Currently there are no studies that evaluate how long it takes for patient's typing skills to return to that of the pre-operative skill level. We would like to answer that question by comparing typing results from different time points including a baseline prior to surgery. We additionally seek to identify which patient characteristics are predictive of a faster return of typing proficiency.

An additional innovative aspect of this project is the use of a web-based typing test that will be used in the assessment of patient typing proficiency. We will additionally use a web-based model for the collection of our survey data.

ELIGIBILITY:
Inclusion Criteria:

* Patients set to undergo carpal tunnel release
* Patients who have a positive EMG test
* Patients must have access to a computer with internet access
* Patients must have an email account
* Patients must be between the ages of 20-70
* Patients that meet typing test requirements

  * Must type weekly
  * Typing proficiency of 30 wpm at time of pre-operative appointment
  * Must use all fingers when typing
  * Can read text in font Times New Roman size 14

Exclusion Criteria:

* People who cannot read or write
* People who do not meet inclusion criteria
* Patients who do not speak English
* Patients unwilling or unable to return for follow-up visits prescribed by the study protocol
* Patients who qualify for inclusion in the study, but refuse to participate.
* Patients with concurrent, ipsilateral confounding hand or upper extremity pathology such as trigger finger, ganglion cyst, painful arthritis, etc.

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Vanderbilt Hand & Upper Extremity Center Outpatient Clinic
Sampling Method: Non-Probability Sample
Enrollment: 38 (Actual)
Dates: Start 2013-05; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Change in typing test measurements (speed and accuracy) | Preoperative, Postoperative: 8-10days, 2wks, 3wks, 4wks, 5wks, 6wks, 8wks, 12wks
  Each patient will complete a preoperative typing test (at their home) prior to undergoing carpal tunnel release surgery. The patient will then take the same typing test at the following time points postoperatively: 8-10days, 2wks, 3wks, 4wks, 5wks, 6wks, 8wks, 12wks. The change in speed and accuracy will be assessed by comparing the preoperative (baseline) typing test results to the postoperative typing test results.

CONTACTS AND LOCATIONS:
Overall Officials: Donald H Lee, MD, Principal Investigator — Vanderbilt University
Locations (1):
- Vanderbilt University Hand & Upper Extremity Center, Nashville, Tennessee, United States